CLINICAL TRIAL: NCT04736732
Title: IRCM Post-COVID-19 (IPCO) Research Clinic: a Multidisciplinary Approach to Evaluate Short and Long-term Complications of COVID-19
Brief Title: Institut de Recherche Cliniques de Montreal (IRCM) Post-COVID-19 (IPCO) Research Clinic
Acronym: IPCO
Status: Recruiting | Type: Observational
Sponsor: Emilia Falcone, MD (Other)
Responsible Party: Sponsor-Investigator, Emilia Falcone, MD, Director, IRCM Post-COVID-19 Research Clinic, Institut de Recherches Cliniques de Montreal
Organization: Institut de Recherches Cliniques de Montreal (Other)
Other Study IDs: 2021-1092
Record Dates: First submitted 2021-02-01; First posted 2021-02-03 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Covid19
Keywords: Post-COVID-19 syndrome; COVID-19-related long-term complications; COVID-19 long haulers; Post-COVID-19 condition; Post-acute sequelae of COVID-19; Long COVID
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva, nasopharyngeal swabs, blood/plasma/serum, peripheral blood mononuclear cells, urine, stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 positive patients: 1. Patients who had previous asymptomatic or mild COVID-19 (mild=never required supplemental oxygen during the acute phase of the infection)
  2. Patients who had previous moderate or severe COVID-19 (moderate=required supplemental oxygen by nasal cannula during the acute phase of the infection; severe=required supplemental oxygen by either high-flow nasal cannula, non-invasive positive pressure ventilation or intubation
  3. Patients who had COVID-19 but did not have signs or symptoms related to COVID-19 lasting beyond 4 weeks from the date of COVID-19 symptom-onset or diagnosis
  Interventions: Other: Medical follow-up
- COVID-19 negative patients: Patients who have not had COVID-19 (i.e., patients who tested negative for COVID-19 and who never had symptoms consistent with COVID-19)
  Interventions: Other: Medical follow-up

INTERVENTIONS:
Other: Medical follow-up — Patients will be followed for medical evaluation and for biobanking of data and biological samples.
  Other Names: Sample collection

SUMMARY:
Sample Size: n=570

Accrual Ceiling: n=627

Study Population: Patients age 18 to 100 years

The study duration includes 51 months to recruit patients and 24 months of total follow-up time counted from the first day of COVID-19 symptoms or date of confirmed COVID-19 diagnosis.

Study Design: This is a prospective, observational cohort study to evaluate the short- and long-term end-organ complications of COVID-19 and to establish a COVID-19 biobank.

Participant Cohorts:

1. Individuals who had previous asymptomatic or mild COVID-19 (mild=never required supplemental oxygen during the acute phase of the infection)
2. Individuals who had previous moderate or severe COVID-19 (moderate=required supplemental oxygen by nasal cannula during the acute phase of the infection; severe=required supplemental oxygen by either high-flow nasal cannula, non-invasive positive pressure ventilation or intubation)
3. Individuals who had COVID-19 but did not have signs or symptoms related to COVID-19 lasting beyond 4 weeks from the date of COVID-19 symptom-onset or diagnosis
4. Individuals who have not had COVID-19 (i.e. individuals who tested negative for COVID-19 and who never had symptoms consistent with COVID-19)

DETAILED DESCRIPTION:
Primary Objectives:

1. Evaluate the short- and long-term end-organ complications post-COVID-19 in relation to the severity of the acute COVID-19 infection.
2. Establish a post-COVID-19 biobank.

Secondary Objectives:

1) Develop a model that may predict the development of end-organ complications.

Primary Endpoint:

The development of any end-organ complication that can plausibly be related to COVID-19.

Secondary Endpoints:

1. Detection of any new abnormality on echocardiogram >4 weeks after COVID-19 symptom-onset or diagnosis.

   Detection of any new abnormality on pulmonary function testing (PFT) or any change in PFT compared to a pre- or post-COVID-19 baseline PFT.
2. An increase in liver enzymes > 2 times upper limit of normal that occurs post-COVID-19 and is not associated to any other process (e.g. cholestasis, drug toxicity, alcohol abuse, hepatitis A, B, C, D, E).
3. Any change in pre-COVID-19 weight, waist circumference or body mass composition.
4. Any change in glycated hemoglobin (HgA1C), lipid profile, thyroid stimulating hormone (TSH), T4 from pre-COVID-19 baseline that begins or persists >4 weeks after COVID-19 symptom-onset or diagnosis.
5. A positive fecal calprotectin or lactoferrin measurement occurring >4 weeks after COVID-19 symptom-onset or diagnosis.
6. Any significant change in renal parameters (e.g. micro-albuminuria, serum creatinine, glomerular filtration rate [GFR]) detected >4 weeks after COVID-19 symptom-onset or diagnosis.
7. Any change in dietary habits (nutritional quantity and quality) as measured by the Food Frequency Questionnaire, in physical activity as measured by actimeter reading, and/or well-being as measured by our Well-Being Questionnaire.

Methodology:

Individuals diagnosed with COVID-19 (for more than 28 days) will have up to 5 medical visits (depending on the time since diagnosis) over the course of 24 months from the date of COVID-19 symptom onset or diagnosis. COVID-19 negative individuals will have up to 3 medical visits. The data will be collected for clinical monitoring and biobanking purposes.

Medical visits include:

* Clinical assessment
* Epidemiological questionnaire
* Well-being questionnaire
* Food frequency questionnaire
* Physical exam (if indicated)
* Vital signs
* Measurement of waist circumference
* Weight and height measurement
* Impedance / evaluation of body mass composition
* Actimeter reading
* Pulmonary function test
* Echocardiography
* Electrocardiogram
* Urine collection
* Blood draw
* Saliva collection
* Stool collection (optional)
* Nasopharyngeal swab (optional)

ELIGIBILITY:
Inclusion Criteria:

* Any gender, ≥ 18 years old
* Current resident of Quebec
* Speaks English or French
* Have a personal email (to which to send reminders and questionnaire by email )

AND

1 of the following criteria:

* At least one COVID-19 positive PCR test, serology or antibody/antigen test in the last 24 months at day of recruitment.
* In the absence of a positive COVID-19 test, the patient had symptoms consistent with COVID-19 while living with a person who had a confirmed positive PCR/serology COVID-19 test.
* Individual who tested negative for COVID-19 while living with a household member who tested positive for COVID-19 (control group), and never had any COVID-19 related symptoms.
* Individual who doesn't have any COVID-19 related symptoms actually, has never had tested positive, and has had at least one negative PCR test.

Exclusion Criteria:

* Any participant not deemed appropriate for enrollment according to the PI
* Known pregnancy (female will not be automatically screened for pregnancy upon enrollment unless there is a possibility that they might be pregnant)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Adults who have had a positive diagnosis of COVID-19.
  * Adults who have tested negative for COVID-19 (control group)
Sampling Method: Non-Probability Sample
Enrollment: 570 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2027-05-04 (Estimated); Study Completion 2027-11-04 (Estimated)

PRIMARY OUTCOMES:
Evaluate the short- and long-term end-organ complications post-COVID-19 in relation to the severity of the acute COVID-19 infection. | 2 years
Establish a post-COVID-19 biobank. | 2 years

SECONDARY OUTCOMES:
The development of any end-organ complication that can plausibly be related to COVID-19. We will evaluate the following end-organ systems: neurological, cardiovascular, pulmonary, renal, endocrine and metabolic, gastro-intestinal (GI). | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Emilia Liana Falcone, M.D., Ph.D., Principal Investigator — IRCM
Locations (1):
- Institut de Recherches Cliniques de Montreal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Future collaborations will be possible with data from the biobank. All data will be anonymous and a committee will evaluate requests for access to the biobank. The principal investigator is responsible for the biobank.
Access Criteria: Recognized researcher collaborating with PI.